CLINICAL TRIAL: NCT01252485
Title: Registry Study on Patient Characteristics, Biological Disease Profile and Clinical Outcome in Acute Myeloid Leukemia and Related Neoplasms - The Biology and Outcome (BiO)-Project
Acronym: AMLSG BiO
Status: Recruiting | Type: Observational
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Prof. Dr. Hartmut Doehner, Prof. Dr., University of Ulm
Other Study IDs: AMLSG BiO
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Acute Myeloid Leukemia (AML); MDS/AML
Keywords: AML; Registry study; Biology and Outcome; MDS/AML
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a registry study in adult patients with newly diagnosed or refractory/relapsed myeloid neoplasms

Investigator's sites: 80-90 sites in Germany and Austria

Estimated duration of observation of an individual patient:

10 years maximum

Objectives

* To register all patients with AML and related neoplasms, newly diagnosed or relapsed/refractory in all AMLSG participating centers (completeness)
* To perform rapid analyses of disease-related genetic markers (incidences, treatment recommendations)
* To assess patient and family history, as well as patient characteristics
* To evaluate treatment response (CR, CRh, CRi) and outcome data (event-free survival [EFS], relapse-free survival [RFS], cumulative incidence of relapse [CIR], cumulative incidence of death [CID], overall survival [OS])
* To evaluate the impact of measurable residual disease (MRD) by different methods
* To assess biological disease features and correlate with clinical outcome data (prognostic and predictive markers)
* To store biosamples from all patients (e.g., bone marrow, blood, plasma, normal tissue; e.g., skin biopsy, finger nails, hairs, sputum, or urine)

ELIGIBILITY:
Inclusion Criteria:

* Patients with suspected diagnosis of acute myeloid leukemia and related neoplasms, newly diagnosed or relapsed/refractory, classified according to the International Consensus Classification
* Age ≥ 18 years. There is no upper age limit.
* Signed written informed consent

Exclusion Criteria:

* Severe neurological or psychiatric disorder interfering with ability to give an informed consent
* No consent for registration, storage and processing of the individual patient and disease characteristics and course as well as information of the family physician about study participation
* No consent for biobanking of patient's biological specimens and performance of analyses on stored material.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with newly diagnosed or relapsed/refractory AML in all AMLSG participating centers (80-90 centers in Germany and Austria)
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2010-07-06 (Actual); Primary Completion 2044-12-31 (Estimated); Study Completion 2044-12-31 (Estimated)

PRIMARY OUTCOMES:
incidence of disease-related genetic markers | 4 weeks
  To perform rapid analyses of disease-related genetic markers (according to International Consensus Classification 2022) (incidences, treatment recommendations)
Event-free survival | 10 years
  To assess patient and family history, patient characteristics and outcome data (event-free survival [EFS], cumulative incidence of relapse [CIR], cumulative incidence of death [CID], overall survival [OS])
Cumulative incidence of relapse | 10 years
  To assess patient and family history, patient characteristics and outcome data (event-free survival [EFS], cumulative incidence of relapse [CIR], cumulative incidence of death [CID], overall survival [OS])
Cumulative incidence of death | 10 years
  To assess patient and family history, patient characteristics and outcome data (event-free survival [EFS], cumulative incidence of relapse [CIR], cumulative incidence of death [CID], overall survival [OS])
Overall survival | 10 years
  To assess patient and family history, patient characteristics and outcome data (event-free survival [EFS], cumulative incidence of relapse [CIR], cumulative incidence of death [CID], overall survival [OS])
Treatment decision (intensive, non-intensive, investigational) | 1 year
  To perform rapid analyses of disease-related genetic markers (according to ICC 2022) (incidences, treatment recommendations)
quality of life | 2 years
  Quality of life assessed by the EORTC Quality of Life Core Questionnaire (QLQ-C30), supplemented by information on self-assessed concomitant diseases, late treatment effects, socioeconomics, and demographics according to Messerer D et al (2008), 6, 12 and 24 months after registration.
Geographical representation | 1 day
  Geographical representation of patients through collection of patients zip codes
Response to therapy | 1 year
  Rate of response: complete remission (CR), CR with partial hematologic recovery (CRh); CR with incomplete hematologic recovery (CRi)
Relapse-free survival | 10 years
Measurable residual disease (MRD) | 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Döhner, Prof. Dr., Study Chair — University Hospital of Ulm
Locations (94):
- Austria (8):
  - Medizinische Universität Graz, Graz
  - Medizinische Universität Innsbruck, Innsbruck
  - Krankenhaus der Barmherzigen Schwestern Linz Betriebsgesellschaft m.b.H., Linz
  - Krankenhaus der Elisabethinen Linz GmbH, Linz
  - Kepler Universitätsklinikum GmbH, Linz
  - Landeskrankenhaus Feldkirch, Rankweil
  - Universitätsklinikum der PMU Landeskrankenhaus Salzburg, Salzburg
  - Hanuschkrankenhaus Wien, Vienna
- Germany (86):
  - Klinikum Aschaffenburg, Aschaffenburg
  - Klinikum Augsburg, Augsburg
  - Ubbo-Emmius-Klinik Aurich, Aurich
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Vivantes Klinikum am Urban, Berlin
  - Vivantes Netzwerk für Gesundheit GmbH Klinikum Neukölln, Berlin
  - Charité Universitätsmedizin Berlin Campus Virchow Klinikum, Berlin
  - Helios Klinikum Emil von Behring, Berlin
  - Vivantes Klinikum Spandau, Berlin
  - Augusta-Kranken-Anstalt, Bochum
  - Medizinische Universitätsklinik Knappschaftskrankenhaus Bochum, Bochum
  - Universitätsklinikum Bonn, Bonn
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Klinikum Bremen-Mitte gGmbH, Bremen
  - Klinikum Darmstadt, Darmstadt
  - St. Johannes Hospital, Dortmund
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - Marien Hospital Düsseldorf GmbH, Düsseldorf
  - Kliniken Essen-Süd Evang. Krankenhaus Essen-Werden gGmbH, Essen
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - St. Franziskus Hospital, Flensburg
  - Städtische Kliniken Frankfurt am Main-Höchst, Frankfurt
  - Medizinische Universitätsklinik, Freiburg im Breisgau
  - MVZ Osthessen Medizinisches Versorgungszentrum, Fulda
  - Klinik der Justus-Liebig-Universität, Giessen
  - Wilhelm-Anton-Hospital gGmbH, Goch
  - Alb Fils Kliniken GmbH, Göppingen
  - Universitätsmedizin Göttingen, Göttingen
  - Universitätsmedizin Greifswald, Greifswald
  - Universitätsklinikum Hall, Halle
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Asklepios Kliniken Hamburg GmbH St. Georg, Hamburg
  - Evangelisches Krankenhaus Hamm, Hamm
  - Klinikum Hanau gGmbH, Hanau
  - Klinikum Hannover Siloah, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Marienhospital Herne Klinikum der Ruhr-Universität Bochum, Herne
  - Universitätsklinikum des Saarlandes, Homburg/Saar
  - Westpfalz-Klinikum Kaiserslautern, Kaiserslautern
  - Städtisches Klinikum Karlsruhe, Karlsruhe
  - St. Vincentius-Kliniken Karlsruhe, Karlsruhe
  - Klinikum Kassel GmbH, Kassel
  - Städtisches Krankenhaus Kiel GmbH, Kiel
  - Helios Klinikum Krefeld, Krefeld
  - Klinikum Landshut gGmbH, Landshut
  - Caritas Krankenhaus Lebach, Lebach
  - Klinikum Lippe-Lemgo, Lemgo
  - Klinikum der Stadt Ludwigshafen am Rhein gGmbH, Ludwigshafen
  - Universitätslinikum Schleswig-Holstein, Lübeck, Lübeck
  - Klinikum Lüdenscheid, Lüdenscheid
  - Univ-Klinikum der Otto-von-Guericke-Universität, Magdeburg
  - Klinikum Magdeburg gGmbH, Magdeburg
  - Universitätsklinikum der Johannes Gutenberg-Universität Mainz, Mainz
  - Klinikum Hochsauerland GmbH, Meschede
  - Johannes Wesling Klinikum Minden, Minden
  - Klinikum Schwäbisch-Gmünd, Mutlangen
  - Evangelisches Krankenhaus Mülheim an der Ruhr GmbH, Mühlheim
  - Klinikum Schwabing, München
  - Klinikum rechts der Isar der TU München, München
  - Städtische Kliniken Neuss Lukaskrankenhaus GmbH, Neuss
  - Sana Klinikum Offenbach, Offenbach
  - Ortenau Klinikum, Offenburg-Gengenbach, Offenburg
  - Pius Hospital Oldenburg, Oldenburg
  - Klinikum Oldenburg gGmbH, Oldenburg
  - Klinikum Passau, Passau
  - Ernst-von-Bergmann-Klinikum Potsdam gGmbH, Potsdam
  - Klinikum Vest, Recklinghausen
  - Universitätsklinikum, Regensburg
  - University hospital Rostock, Rostock
  - Akademisches Lehrkrankenhaus des Saarlandes St. Theresia, Saarbrücken
  - Marienhaus Klinikum St. Elisaeth Saarlouis, Saarlouis
  - Nordwest-Krankenhaus Sanderbusch, Sande
  - Klinikum Stuttgart Katharinenhospital, Stuttgart
  - Diakonie-Klinikum Stuttgart, Stuttgart
  - Vinzenz von Paul Kliniken gGmbH Marienhospital Stuttgart, Stuttgart
  - Klinikum Traunstein, Traunstein
  - Klinikum Mutterhaus der Borromäerinnen gGmbH, Trier
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Medizinische Universitätsklinik Tübingen, Tübingen
  - University Hospital of Ulm, Ulm
  - Universitätsklinik Ulm Labor für Zytogenetische und Molekulare Diagnostik, Ulm
  - Schwarzwald-Baar Klinikum Villingen-Schwenningen GmbH, Villingen-Schwenningen
  - Harzklinikum Dorothea Christiane Erxleben, Wernigerode
  - Helios Klinikum Wuppertal, Wuppertal